CLINICAL TRIAL: NCT02906267
Title: Ultrasonographic Comparison of Gastric Volume After Three Modes of Positive Facemask. A Prospective Randomized Study.
Brief Title: Ultrasonographic Comparison of Gastric Volume After Three Modes of Positive Facemask During Induction of Anaesthesia
Acronym: UGV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Principal Investigator, LAFERE Pierre, Docteur Pierre Lafère, University Hospital, Brest
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Ultrasonic gastric volume
Record Dates: First submitted 2016-09-05; First posted 2016-09-20 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Positive-Pressure Respiration; Respiratory Aspiration of Gastric Content

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Manual-controlled (Other): Patient in the manual ventilation group will receive facemask ventilation to get a tidal volume of 8-10ml/kg with a respiratory rate of 15/min. The pop-off valve will be set to 20 cm H2O.
  Interventions: Other: Diagnostic ultrasonography of gastric volume
- Volume-controlled (Other): mechanical breath will be delivered by a Primus ventilator (Dräger, Lubeck, Germany) at a frequency of 15 breath/min. Tidal volume will be set to 8-10 ml/min.
  Interventions: Other: Diagnostic ultrasonography of gastric volume
- Pressure-controlled (Other): mechanical breath will be delivered by a Primus ventilator (Dräger, Lubeck, Germany) at a frequency of 15 breath/min. Pressure will be adjusted to obtain a tidal volume of 8-10 ml/min.
  Interventions: Other: Diagnostic ultrasonography of gastric volume

INTERVENTIONS:
Other: Diagnostic ultrasonography of gastric volume — Ultrasonic measurement of gastric insufflation during positive pressure ventilation (secondary endpoint) and final gastric volume after positive pressure ventilation (primary endpoint)

SUMMARY:
This study is designed to evaluate the occurrence of gastric insufflation and the critical volume of the stomach after three different modes of positive pressure ventilation during induction (Manual-controlled, volume-controlled and pressure-controlled ventilation)

DETAILED DESCRIPTION:
Aspiration of gastric contents can be a serious perioperative complication, which can be related to facemask positive pressure ventilation with unprotected airway. Even with low peak airway pressure (<15 cm H2O) gastric insufflation may occur. Since gastric content and volume assessment is a new point-of-care ultrasound recommended application, the cross-sectional antra area will be measured using ultrasonography before, continuously during facemask ventilation and after intubation.

ELIGIBILITY:
Inclusion Criteria:

* ASA status I and II

Exclusion Criteria:

* Pregnant woman Obese patient (BMI>30kgm-2) oropharyngeal or facial anomalies anticipated difficult mask ventilation upper respiratory tract infection history of gastric surgery patient refusal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Gastric volume before and after positive pressure ventilation | 15 minutes

SECONDARY OUTCOMES:
Ultrasonographic detection of gastric insufflation during ventilation | 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Pierre LAFERE, MD,PhD, Principal Investigator — CHRU de Brest
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Undecided